CLINICAL TRIAL: NCT01289080
Title: A Single-dose, Open-label, Parallel-group, Matched Trial Evaluating the Pharmacokinetics of Oral OPC-34712 Tablets in Subjects With Normal Renal Function and Renally Impaired Subjects
Brief Title: Trial Evaluating OPC-34712 in Subjects With Normal Renal Function and Renally Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 331-09-226
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia; Psychiatric Disorders
Keywords: Schizophrenia; psychiatric disorders; renal failure
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): subjects with normal renal function
  Interventions: Drug: OPC-34712
- Group 2 (Active Comparator): severely renally impaired subjects
  Interventions: Drug: OPC-34712

INTERVENTIONS:
Drug: OPC-34712 — administered orally

SUMMARY:
This trial is an open-label, multi-center, parallel-arm, single-dose trial in 2 groups: 1 group of subjects with normal renal function and 1 group of severely renally impaired subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (non-childbearing potential) subjects ≥ 18 years of age.
* Ability to provide written informed consent prior to initiation of any trial-related procedures, and ability, in the opinion of the principal investigator, to comply with all the requirements of the trial.
* Male and female subjects who are surgically sterile; female subjects who have been postmenopausal for at least 12 consecutive months (confirmed by follicle stimulating hormone sample at Screening); or male subjects who agree to remain abstinent or to practice double-barrier forms of birth control and refrain from sperm donation from trial Screening through 90 days from the last dose of the investigational medicinal product.
* Body weight within ± 35% of ideal body weight as defined in the 1983 Metropolitan Height and Weight Tables (see Appendix 4, Appendix 5, and Appendix 6). Minimum body weight no less than 50 kg.

Inclusion Criteria for Subjects with Normal Renal Function

* Subjects who are in good health as determined by a medical history, physical examination, serum chemistry, hematology, urinalysis, hepatitis B and C tests, and human immunodeficiency virus (HIV) testing.
* Creatinine clearance > 80 mL/min indicating normal renal function.

Inclusion Criteria for Renally Impaired Subjects

* Renally impaired subjects may be taking medications which, in the opinion of the clinical investigator and sponsor, are believed to be therapeutic for the subjects (but do not affect OPC-34712 absorption, distribution, metabolism, or elimination). Inhibitors and inducers of CYP3A4 and inhibitors of CYP2D6 are not allowed.
* Creatinine clearance < 30 mL/min indicating severe renal impairment.
* Subjects with renal impairment should have relatively stable renal function as determined by creatinine clearance and otherwise be in generally good health.

Exclusion Criteria:

Clinically significant abnormality in past medical history, or at the screening physical examination, that in the investigator's or sponsor's opinion may place the subject at risk or interfere with outcome variables including absorption, distribution, metabolism, and excretion of drug.

* Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion, or any other condition that may place the subject at risk.
* History of drug and/or alcohol abuse within 2 years prior to Screening.
* A positive urine alcohol test and/or urine drug screen for substance of abuse at Screening or upon check-in to the trial site.
* The donation of blood or plasma within 30 days prior to dosing.
* Any history of significant bleeding or hemorrhagic tendencies.
* History of or current hepatitis or carriers of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibodies (anti-HCV).
* History of acquired immunodeficiency syndrome or determined human immunodeficiency virus (HIV) positive at Screening.
* Use of an investigational drug or product, or participation in a drug trial within 30 days prior to dosing.
* Previous exposure to OPC-34712.
* History of clinically significant drug allergies or sensitivities.
* Subjects who are pregnant or breastfeeding. A negative serum pregnancy test must be confirmed prior to administration of trial medication for all female subjects.
* Subjects who have a supine pulse rate, after resting for ≥ 3 minutes, outside the range of 40 to 90 bpm. The sponsor may allow exceptions if they are not deemed clinically significant.

Exclusion Criteria for Healthy Subjects

* Clinically significant abnormal findings in the serum chemistry, hematology, or urinalysis results obtained at Screening or Day -1.
* Use of prescription, over-the-counter, herbal medication or vitamin supplements within 14 days prior to dosing and antibiotics within 30 days prior to dosing. The sponsor may allow exceptions only if the medication's administration is deemed unlikely to impact the pharmacokinetic result. Inhibitors and inducers of CYP3A4 and inhibitors of CYP2D6 are not allowed.
* Subjects who have supine, sitting, or standing blood pressure, after resting for ≥ 3 minutes, higher than 130/80 mmHg or lower than 100/50 mmHg. The sponsor may allow exceptions if they are not deemed clinically significant.

Exclusion Criteria for Renally Impaired Subjects

* Subjects that have undergone a renal transplant.
* Renally impaired subjects may be taking medications which, in the opinion of the clinical investigator and sponsor, are believed to be therapeutic for the subjects (but do not affect OPC-34712 absorption, distribution, metabolism, or elimination). Inhibitors and inducers of CYP3A4 and inhibitors of CYP2D6 are not allowed.
* Clinically significant abnormal findings in the serum chemistry, hematology, or urinalysis results obtained at Screening or Day -1, other than those associated with underlying renal conditions and other stable medical conditions consistent with the disease processes.
* Subject requiring dialysis or expected to require dialysis within 45 days.
* Subjects who have supine, sitting, or standing blood pressure, after resting for ≥ 3 minutes, higher than 160/95 mmHg or lower than 100/50 mmHg. The sponsor may allow exceptions if they are not deemed clinically significant.
* Subjects with evidence of delirium.
* Clinically relevant changes on electrocardiogram such as any atrioventricular block, prolongation of the QRS complex over 120 msec (for both male and female subjects), or with a QTcF interval ≥ 450 msec.
* Any subject who, in the opinion of the sponsor or the investigator, should not participate in the trial.
* Consumption of alcohol and/or food and beverages containing methylxanthines, grapefruit, grapefruit juice, Seville oranges, or Seville orange juice within 72 hours prior to dosing.
* Use of any drug known or suspected of inhibiting or stimulating hepatic drug metabolism enzymes within 30 days prior to Screening.
* Exposure to any substances known to stimulate hepatic microsomal enzymes within 30 days prior to Screening through the end of the trial (eg, occupational exposure to pesticides, organic solvents).
* History of serious mental disorders.
* Major surgery of the digestive tract (excluding appendectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Skuban, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (2):
- United States (2):
  - Otsuka Investigational Site, Miami, Florida
  - Otsuka Investigational Site, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was an open-label, multicenter, parallel-arm, single-dose trial in two groups: 1 group of participants with normal renal function and 1 group of severely renally impaired participants.
Pre-assignment Details: The participant assignment was made based on Urine Creatinine Clearance (urine CLcr). If the urine CLcr was < 30 mL/minute for renally impaired participants and the urine CLcr was > 80 mL/minute for participants with normal renal function.
Groups:
- Normal: Participants with normal renal function were administered 3 mg brexpiprazole on Day 1.
- Renally Impaired: Participants with severe renal impairment were administered 3 mg brexpiprazole on Day 1.
Period: Overall Study
Arm/Group | Normal | Renally Impaired
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal | Renally Impaired | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (10.1) | 62.9 (12.2) | 60.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Unbound Area Under the Concentration (AUC) Time Curve Calculated to the Last Observable Concentration Brexpiprazole (AUCt,u).
Description: Blood samples were collected on Day 1 at Predose (within 15 minutes of dosing) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours Postdose or at Early Termination (ET). Unbound fraction of drug in plasma was calculated as 100% - mean percent of brexpiprazole bound to plasma protein for each participant.
Time Frame: Day 1 to Day 8
Population: The dataset for pharmacokinetics (PK) analysis of all evaluable brexpiprazole PK parameters consisted of enrolled participants who had evaluable plasma concentrations.
Measure: Mean (Standard Deviation); unit: nanograms*hours/mL (ng*h/mL)
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 9 | 10
nanograms*hours/mL (ng*h/mL) | 8.17 (1.37) | 13.3 (6.26)

2. Primary Outcome: Unbound Area Under AUC- Time Curve From Time Zero to Infinity (AUC∞,u).
Description: Blood samples were collected at Predose (within 15 minutes of dosing) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours or at ET. Unbound fraction of drug in plasma was calculated as 100% - mean percent of brexpiprazole bound to plasma protein for each participant.
Time Frame: Day 1 to Day 8
Population: The dataset for PK analysis of all evaluable brexpiprazole PK parameters consisted of enrolled participants who had evaluable plasma concentrations.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Renally Impaired: Participants with severe renal impairment were administered 3 mg brexpiprazole Day 1.
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 7 | 7
ng*h/mL | 9.58 (2.26) | 18.0 (8.72)

3. Primary Outcome: Unbound Maximum (Peak) Plasma Concentration of Brexpiprazole (Cmax,u).
Description: as for outcome 2
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 9 | 10
ng/mL | 0.195 (0.0662) | 0.198 (0.0702)

4. Secondary Outcome: AUC Time Curve of Brexpiprazole Metabolite (DM-3411) Calculated to the Last Observable Concentration at Time t (AUCt).
Description: Blood samples were collected at Predose (within 15 minutes of dosing) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours or at ET. The AUCt was estimated using the linear trapezoidal rule.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 9 | 9
ng*h/mL | 1410 (423) | 2080 (1230)

5. Secondary Outcome: AUC Time Curve of Brexpiprazole From Time Zero to Infinity (AUC∞).
Description: Blood samples were collected at Predose (within 15 minutes of dosing) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours or at ET. The AUC∞ was estimated using the linear trapezoidal rule.
Time Frame: Day 1 to Day 8
Population: The dataset for PK analysis of all evaluable brexpiprazole PK parameters consisted of enrolled participants who had evaluable plasma concentrations. AUC-time curve from zero to infinity (AUC∞) was not determined for DM-3411 metabolite.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 7 | 7
ng*h/mL | 2050 (510) | 3800 (1970)

6. Secondary Outcome: Maximum Plasma Concentration of Brexpiprazole Metabolite (DM-3411) (Cmax).
Description: as for outcome 2
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 9 | 10
ng/mL | 18.2 (6.24) | 19.8 (12.3)

7. Secondary Outcome: Time to Cmax of Brexiprazole Metabolite (DM-3411) (Tmax).
Description: Blood samples were collected at Predose (within 15 minutes of dosing) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours or at ET. Tmax is the time taken to reach highest measured concentration of the drug during the dosing interval.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 9 | 10
h | 12.0 (1.00-8.00) [8.00 to 24.00] | 30.0 (2.00-8.00) [3.00 to 144]

8. Secondary Outcome: Apparent Clearance From Plasma After Extravascular Administration of Brexpiprazole (CL/F).
Description: The value of CL/F was determined as Dose/AUC∞. Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) was influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance was a quantitative measure of the rate at which a drug substance was removed from the blood.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 7 | 7
mL/h/kg | 23.0 (8.05) | 14.2 (6.46)

9. Secondary Outcome: Unbound Fraction of Brexpiprazole in Plasma (fu).
Description: as for outcome 2
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of unbound brexpiprazole in plasma
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 9 | 10
% of unbound brexpiprazole in plasma | 0.476 (0.0525) | 0.492 (0.0346)

10. Secondary Outcome: Apparent Unbound Clearance From Plasma After Extravascular Administration of Brexpiprazole (CLu/F).
Description: as for outcome 2
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 7 | 7
mL/h/kg | 0.110 (0.0493) | 0.0686 (0.0336)

11. Secondary Outcome: Terminal-phase Elimination Half-life of Brexpiprazole (t1/2,z).
Description: as for outcome 2
Time Frame: Day 1 to Day 8
Population: The dataset for PK analysis of all evaluable brexpiprazole PK parameters consisted of enrolled participants who had evaluable plasma concentrations. The terminal phase elimination half-life was not determined for DM-3411 metabolite.
Measure: Mean (Standard Deviation); unit: h
Groups:
- Renally Impaired: Participants with severe renal impairement were administered 3 mg brexpiprazole on Day 1.
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 7 | 7
h | 71.7 (23.8) | 87.4 (28.9)

12. Secondary Outcome: Renal Clearance (CLr) of Brexipiprazole Metabolite (DM-3411).
Description: Urine samples were collected at Predose at intervals of 0 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120, 120 to 144, and 144 to 168 hours postdose. Unbound fraction of drug in plasma was calculated as 100% - mean percent of brexpiprazole bound to plasma protein for each participant.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 9 | 9
mL/h/kg | 1.38 (0.883) | 0.683 (0.471)

13. Secondary Outcome: Fraction of the Systemically Available Brexpiprazole Metabolite (DM-3411) Excreted Into the Urine (fe,u).
Description: Urine samples were collected at Predose and at intervals of 0 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120, 120 to 144, and 144 to 168 hours postdose. Unbound fraction of drug in plasma was calculated as 100% - mean percent of brexpiprazole bound to plasma protein for each participant.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of unbound brexpiprazole in urine.
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 9 | 9
% of unbound brexpiprazole in urine. | 3.91 (1.66) | 2.55 (1.19)

14. Secondary Outcome: The Abnormalities Found in Vital Signs, ECGs, and Clinical Laboratory Tests Are Reported as AEs Upon Study Physicians Discretion.
Description: An adverse event (AE) was an exacerbation of an existing problem or any new problem, experienced by a participant when enrolled in a trial, whether or not it was considered drug related by the study physician.
Time Frame: AEs were recorded from Screening (ICF was signed) to Follow-up 31 (+ 2) days.
Population: The dataset for all safety analyses consisted of the data from all enrolled participants who received at least 1 dose of study medication, regardless of any protocol deviation. All observed data for these subjects were included.
Measure: Number; unit: participants
Arm/Group | Normal | Renally Impaired
Number analyzed (Participants) | 9 | 10
participants
  Participants with adverse events | 3 | 5
  Participants with TEAEs | 3 | 5
  Participants with severe TEAEs | 0 | 1

ADVERSE EVENTS:
Time Frame: AEs were recorded from Screening (ICF was signed) to Follow-up 31 (+ 2) days.
Description: A SAE was any untoward medical occurrence that results in death or was life-threatening or required inpatient hospitalization or prolonged hospitalization. An AE was an exacerbation of an existing problem or any new problem, experienced by a participant when enrolled in a trial, whether or not it was considered drug related by the study physician.
Groups:
- Brexpiprazole 3mg: Participants with normal renal function and severe renal impairment were administered 3 mg brexpiprazole.
Arm/Group | Brexpiprazole 3mg
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 8/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 3mg (N=19)
Constipation (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypotension (Vascular disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Orthostatic hypotension (Vascular disorders) | 2
Somnolence (Nervous system disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No